CLINICAL TRIAL: NCT04601116
Title: A Randomized, Multicenter, Double-blind, Placebo-controlled Comparison of Standard (Neo)Adjuvant Therapy Plus Placebo Versus Standard (Neo)Adjuvant Therapy Plus Atorvastatin in Patients With Early Breast Cancer
Brief Title: The MASTER Study (MAmmary Cancer STatin ER Positive Study)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Hospital of Southern Jutland (Other); University of Copenhagen (Other); Bornholms Hospital (Unknown); Naestved Hospital (Other); Vejle Hospital (Other); Odense University Hospital (Other); Nordsjaellands Hospital (Other); Aalborg University Hospital (Other); Herning Hospital (Other)
Responsible Party: Principal Investigator, Signe Borgquist, MD, PhD, Chair Professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBMASTER; 2019-002508-42 (EudraCT Number)
Record Dates: First submitted 2019-07-25; First posted 2020-10-23 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer Female; Estrogen Receptor Positive Tumor
Keywords: Breast Cancer; Atorvastatin; Estrogen Receptor Positiv Tumor; Adjuvant therapy; Neoadjuvant; Statin
MeSH Terms: conditions — Breast Neoplasms | interventions — Atorvastatin; Tablets

STUDY DESIGN:
Intervention Model Description: A prospective, two-armed, randomized (1:1), multicenter, national, double-blind, placebo-controlled study in early breast cancer patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Atorvastatin 80 Mg Oral Tablet (Active Comparator): Atorvastatin 80 mg tablets per day for 2 years
  Interventions: Drug: Atorvastatin 80 Mg Oral Tablet
- Placebo (Placebo Comparator): Placebo tablets 1 per day for 2 years.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Atorvastatin 80 Mg Oral Tablet — Atorvastatin 80 mg per day for 2 years
  Arms: Atorvastatin 80 Mg Oral Tablet
Drug: Placebo oral tablet — Placebo 1 tablet per day for 2 years
  Arms: Placebo

SUMMARY:
Given the compelling evidence supporting a protective effect of statins on breast cancer recurrence, calls for prospective clinical trials have been expressed. In this trial - the MASTER trial - we hypothesize that the addition of statin treatment to the current breast cancer treatment will improve the prognosis of women with early breast cancer. This trial is designed as follows: a randomized, multicenter, double-blind, placebo-controlled comparison of standard (neo)adjuvant therapy plus placebo versus standard (neo)adjuvant therapy plus atorvastatin in patients with early breast cancer.

DETAILED DESCRIPTION:
Cholesterol-lowering drugs such as statins are currently used to lower cholesterol levels and prevent cardiovascular events. Statins have, however, received substantial scientific attention as cancer-inhibiting drugs. Previous findings were recently supported in a large-scaled study again demonstrating the beneficial effects of statins on breast cancer outcome this time nested within a large, international, randomized clinical trial of modern adjuvant cancer therapy. Given the compelling evidence supporting a protective effect of statins on breast cancer recurrence, calls for prospective clinical trials have been expressed. In this trial - the MASTER trial - we hypothesize that the addition of statin treatment to the current breast cancer treatment will improve the prognosis of women with early breast cancer. Thus, the primary objective of the MASTER trial is to determine the clinical efficacy of the statin - atorvastatin - as measured by invasive disease-free survival among patients with primary breast cancer.

The trial is nationwide throughout Denmark and a total of 3,360 women are to be included in the trial. Women eligible for the trial have been diagnosed with an estrogen receptor positive breast cancer and are candidates for systemic cancer therapy, either prior to or following breast surgery. Upon eligibility and signed informed consent, trial participants will be randomized in a 1:1 manner to either standard treatment and atorvastatin 80 mg/day or standard treatment and placebo. The randomization is blinded. The treatment with atorvastatin or placebo will continue for two years unless side effects are experienced and further treatment with atorvastatin or the placebo is deemed inadequate. The standard treatment will of course continue as planned. The trial participants will follow the standard clinical routines in terms of follow-up and in addition they are asked to fill in questionnaires, i.e. regarding potential side effects or new events or diagnoses, up to ten years following inclusion. Potential breast cancer recurrences are hereby identified and a follow-up of at least 61/2 years will be required for the trial the demonstrate the estimated clinical difference between the randomized groups of patients.

ELIGIBILITY:
Patients must meet ALL of the following criteria to be eligible for randomization:

Inclusion Criteria:

1. Women with estrogen receptor positive breast cancer who are candidates for (neo)adjuvant systemic therapy OR have received ≤3 years of adjuvant endocrine therapy.
2. Age > 18 years.
3. Performance status of ECOG ≤ 2.
4. Prior to patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations.

Patients meeting ANY one of the following criteria are not eligible:

Exclusion Criteria:

1. History of any prior (ipsi- and/or contralateral) invasive breast carcinoma.
2. Ongoing (prevalent) cholesterol-lowering therapy (statins, fibrates, ezetimibe, PCSK9 inhibitors). If so, the patient can be enrolled in the observational arm.
3. Evidence of hepatic dysfunction (alanine aminotransferase level more than three times the upper limit of the normal range) or renal dysfunction (creatinine level more than three times the upper limit of the normal range).
4. Predisposing factors for rhabdomyolysis, including hypothyroidism, reduced renal function, any muscle - or liver disease, or excessive alcohol consumption AND creatine kinase (CK) measured to less than five times the upper limit (CK only measured in case of predisposing factors).
5. No current medication with potent CYP3A4-inhibitors (e.g. ketokonazole, erythromycin) or gemfibrozile, cyclosporin or danazol.
6. Pregnancy or breast-feeding.
7. Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; these conditions will be discussed with the patient before registration in the trial.
8. History of allergic reactions attributed to compounds of similar chemical or biological composition to atorvastatin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3360 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Invasive disease-free survival | 10 years
  Invasive disease-free survival (IDFS), defined as the time from randomization until the date of the first occurrence of one of the following events:
  * Ipsilateral invasive breast tumor recurrence: invasive breast cancer involving the same breast parenchyma as the original primary.
  * Regional invasive breast cancer recurrence: Invasive breast cancer in the axilla, regional lymph nodes, chest wall, and skin of the ipsilateral breast.
  * Distant recurrence: Metastatic disease-breast cancer that has either been biopsy confirmed or clinically diagnosed as recurrent invasive breast cancer.
  * Death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause.
  * Contralateral invasive breast cancer.
  * Second primary non-breast invasive cancer.

SECONDARY OUTCOMES:
Distant-recurrence free interval | 10 years
  Distant-recurrence free interval defined as time from inclusion to first distant recurrence including associations with first site of recurrence.
Recurrence-free interval | 10 years
  Recurrence-free interval including associations with first site of recurrence
Overall survival. | 10 years
  Overall survival.
Incidence of Treatment-Emergent Adverse Events as assessed by CTC-AE, 5.0 | 10 years
  Incidence of Treatment-Emergent Adverse Events as assessed by CTC-AE, 5.0
Cardiac death-free interval | 10 years
  Cardiac death-free interval. Cardiac death is defined as:
  1. Definitive cardiac death due to heart failure, myocardial infarction or documented primary arrhythmia.
  2. Probable cardiac death: Probable cardiac death defined as sudden, unexpected death within 24 hours of a definite or probable cardiac event (e.g., syncope, cardiac arrest, chest pain, infarction, arrhythmia) without documented etiology.
Co-morbidity | 10 years
  Co-morbidity incidence beyond cardiovascular events during follow-up including diagnoses such as diabetes mellitus.

CONTACTS AND LOCATIONS:
Overall Officials: Signe SB Borgquist, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospitak, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No